CLINICAL TRIAL: NCT03951584
Title: Prognosis of Vestibular Dysfunction in Patients With Idiopathic Sudden Sensorineural Hearing Loss
Status: Completed | Type: Observational
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: Cohort ISSNHL with vertigo
Record Dates: First submitted 2019-05-06; First posted 2019-05-15 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2020-02

CONDITIONS: Vestibular Disorder; Sudden Hearing Loss
Keywords: idiopathic sudden sensorineural hearing loss; vestibular dysfunction
MeSH Terms: conditions — Vestibular Diseases; Hearing Loss, Sudden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ISSNHL with vertigo: Participants who suffered from ISSNHL with vertigo will be included in this study cohort. Participants will undergo vestibular function tests including caloric test, sensory organization test, video head impulse test and vestibular evoked myogenic potentials at baseline and 2 months after onset, to evaluate the damage and prognosis of vestibular function.
  Interventions: Other: ISSNHL with vertigo

INTERVENTIONS:
Other: ISSNHL with vertigo — Participants who suffered from ISSNHL with vertigo will be included in this study. Participants will undergo vestibular function tests including caloric test, sensory organization test, video head impulse test and vestibular evoked myogenic potentials at baseline and 2 months after onset as primary outcome, to evaluate the damage and prognosis of vestibular function.

SUMMARY:
Idiopathic sudden sensorineural hearing loss (ISSNHL) refers to idiopathic sensorineural hearing loss of at least 30 dB over at least three test frequencies occurring over a 72-hour period. Vertigo has been considered a risk factor of poor prognosis in patients with ISSNHL. However, the clinical outcome and development of vestibular function in these patients have not been reported yet. We'd like to conduct a study on the problem whether these patients resulted in a complete recovery of the peripheral vestibular functions or compensation of the central vestibular system. If the answer is the former one, these cases might be supportive evidence of regeneration of hair cells in vestibular disorders.

DETAILED DESCRIPTION:
This study is designed as a prospective cohort study with only one cohort. Enrolment and data collection are performed by trained research staff who are not involved in the care of the patients. The primary measurement is the vestibular function tests including SOT, the caloric reflex test, vHIT, VEMP (cVEMP and oVEMP). The secondary measurements included PTA, DHI, and VAS. The sample size was set at 60 patients. The continuous variables were expressed as means ± standard deviation (SD) whereas categorical variables were expressed as frequency and percentage for data description. P <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 16 to 70 years old.
* Diagnosed as ISSNHL.
* Present with vertigo.
* At least 1 abnormal result in vestibular function tests(SOT, vHIT, caloric reflex test, and VEMP).
* The onset of the disease was within 30 days.

Exclusion Criteria:

* Unwilling to sign informed consent.
* The cause of sudden hearing loss has been identified, such as trauma, vasogenic disease, et al.
* Bilateral hearing loss.
* Patients with coexisting vestibular disorders, including Meniere disease, vestibular neuritis, labyrinthitis, and peripheral vestibular loss et al.
* Patients not suitable to receiving vestibular function tests, such as those with severe cervical spine disease, cardiovascular disease, or pregnancy et al.
* Cognitive impairment;
* Other conditions that the investigator evaluated the patients as not appropriate for this study.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who suffered from ISSNHL with vertigo and the onset of this disease was within 30 days, will be included in this study cohort. The enrollment of the participants will be held in the clinic of Eye and ENT Hospital of Fudan University.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Abnormal rate of vestibular function in the Sensory Organization Test(SOT) at baseline. | Baseline
  abnormal rate=(number of participants who have abnormal results in vestibular function in SOT at the baseline)/(number of participants in total)
Recovery rate of vestibular input in the Sensory Organization Test(SOT) at 2-months follow-up after onset. | 2 months after onset
  recovery rate=(number of participants who had abnormal results in vestibular function in SOT at the baseline and get normal vestibular function results in SOT at 2-months follow-up after onset)/(number of participants who had abnormal vestibular function results in SOT at the baseline)
Abnormal rate of the caloric test at baseline. | Baseline
  Abnormal rate=(number of participants who have abnormal results in the caloric test at the baseline)/(number of participants in total).
  An abnormal result is considered if unilateral reaction weakening is greater than 22%, and/or directional preponderance is greater than 27%.
Recovery rate of the caloric test at 2-months follow-up after onset. | 2 months after onset
  recovery rate=(number of participants who had abnormal results in the caloric test at the baseline and get normal results in the caloric test at 2-months follow-up after onset)/(number of participants who get abnormal results in the caloric test at the baseline).
  An abnormal result is considered if unilateral reaction weakening is greater than 22%, and/or directional preponderance is greater than 27%.
Abnormal rate of the vHIT at baseline. | Baseline
  Abnormal rate=(number of participants who have abnormal results in vHIT at the baseline)/(number of participants in total).
  An abnormal result is considered if there are pathological saccades and the gain of each semicircular canal is out of normal range.
Recovery rate of the vHIT at 2-months follow-up after onset. | 2 months after onset
  recovery rate=(number of the participants who had abnormal results in vHIT at the baseline and get normal results in vHIT at 2-months follow-up after onset)/(number of the participants who get abnormal results in vHIT at the baseline).
  An abnormal result is considered if there are pathological saccades and the gain of each semicircular canal is out of normal range.
Abnormal rate of Cervical Vestibular Evoked Myogenic Potentials (cVEMP) at baseline. | Baseline
  Abnormal rate=(number of participants who have abnormal results in cVEMP at the baseline)/(number of participants in total) The abnormal result is considered if potentials were not elicited or out of normal range, or the asymmetrical ratio is larger than normal.
Recovery rate of Cervical Vestibular Evoked Myogenic Potentials (cVEMP) at 2-months follow-up after onset. | 2 months after onset
  recovery rate=(number of the participants who had abnormal results in cVEMP at the baseline and get normal results in cVEMP at 2-months follow-up after onset)/(number of the participants who had abnormal results in cVEMP at the baseline) The abnormal result is considered if potentials were not elicited or out of normal range, or the asymmetrical ratio is larger than normal.
Abnormal rate of Ocular Vestibular Evoked Myogenic Potentials (oVEMP) at baseline. | Baseline
  Abnormal rate=(number of participants who had abnormal results in oVEMP at the baseline)/(number of participants in total) The abnormal result is considered if potentials were not elicited or out of normal range, or the asymmetrical ratio is larger than normal.
Recovery rate of Ocular Vestibular Evoked Myogenic Potentials (oVEMP) at 2-months follow-up after onset. | 2 months after onset
  recovery rate=(number of the participants who had abnormal results in oVEMP at the baseline and get normal results in oVEMP at 2-months follow-up after onset)/(number of the participants who had abnormal results in oVEMP at the baseline) The abnormal result is considered if potentials were not elicited or out of normal range, or the asymmetrical ratio is larger than normal.

SECONDARY OUTCOMES:
Change of Dizziness Handicap Inventory at 2 months after onset | 2 months after onset
  Mean value of change of DHI from baseline at 2 months after onset in each participant.
  Subjective evaluation of vertigo by participants. Score range from 0 to 100 (0 refers to no influence on daily life, while 100 refers to the most severe influence on patient's daily life.)
Change of Visual Analogue Scale in Vertigo at 2 month after onset | 2 months after onset
  Mean value of change of VAS-V from baseline at 2 months after onset in each participant.
  Subjective evaluation of vertigo by participants. Score from 0 to 10. The larger the score, the more severe the vertigo is.
Change of Pure Tone Audiometry(PTA) at 2 months after onset | 2 months after onset
  mean value of change of PTA in each participant at 2 months after onset from baseline (if the participants can provide with an earlier PTA result before enrollment and after onset, which we believe is of high possibility, this PTA result will be considered as baseline parameters).

CONTACTS AND LOCATIONS:
Overall Officials: Huawei Li, Phd & MD, Study Chair — Eye and ENT Hospital of Fudan University
Locations (1):
- Otorhinolaryngology Department of Affiliated Eye and ENT Hospital, Fudan University, Shanghai, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
For IPD please contact the author at haoweiming1993@163.com
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Stachler RJ, Chandrasekhar SS, Archer SM, Rosenfeld RM, Schwartz SR, Barrs DM, Brown SR, Fife TD, Ford P, Ganiats TG, Hollingsworth DB, Lewandowski CA, Montano JJ, Saunders JE, Tucci DL, Valente M, Warren BE, Yaremchuk KL, Robertson PJ; American Academy of Otolaryngology-Head and Neck Surgery. Clinical practice guideline: sudden hearing loss. Otolaryngol Head Neck Surg. 2012 Mar;146(3 Suppl):S1-35. doi: 10.1177/0194599812436449. PMID 22383545
- [Background] Wen YH, Chen PR, Wu HP. Prognostic factors of profound idiopathic sudden sensorineural hearing loss. Eur Arch Otorhinolaryngol. 2014 Jun;271(6):1423-9. doi: 10.1007/s00405-013-2593-y. Epub 2013 Jun 15. PMID 23771280
- [Background] Yu H, Li H. Association of Vertigo With Hearing Outcomes in Patients With Sudden Sensorineural Hearing Loss: A Systematic Review and Meta-analysis. JAMA Otolaryngol Head Neck Surg. 2018 Aug 1;144(8):677-683. doi: 10.1001/jamaoto.2018.0648. PMID 29931169
- [Background] Rauch SD. Clinical practice. Idiopathic sudden sensorineural hearing loss. N Engl J Med. 2008 Aug 21;359(8):833-40. doi: 10.1056/NEJMcp0802129. No abstract available. PMID 18716300
- [Derived] Hao W, Ye L, Yu H, Li H. Prognosis of vestibular dysfunction in idiopathic sudden sensorineural hearing loss with vertigo: a prospective cohort study. J Neurol. 2023 Nov;270(11):5516-5526. doi: 10.1007/s00415-023-11894-w. Epub 2023 Jul 30. PMID 37517037